CLINICAL TRIAL: NCT06102187
Title: Fujian Cohort Study of cARdiomEtabolic Disease and Comorbidity(Fu-CARE)
Brief Title: Cohort Study in Fujian Province
Status: Recruiting | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Collaborators: Center for Disease Control and Prevention, Fujian (Other); China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Kaiyang Lin, Deputy director, Fujian Provincial Hospital
Other Study IDs: LYu
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Chronic Disease
Keywords: Cardiovascular and metabolic disease comorbidity
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Urine samples for biochemical tests, biomarker examination and DNA extraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, Chinese residents aged 35 to 75 years old were recruited from Fujian Province. Physical examination, questionnaire survey and biological sample collection were performed at baseline, and at least 4 years of follow-up were conducted. Information on newly discovered cardiovascular metabolic illnesses and comorbidities was collected during follow-up, and repeated surveys similar to baseline were conducted. To explore the relationship between environment, diet and lifestyle and the risk of cardiovascular metabolic diseases and concomitant disorders.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-75, having lived in Fuzhou, Putian, Quanzhou, Nanping, Xiamen, Zhangzhou, Longyan, Sanming, or Ningde in Fujian Province for more than 6 months.

Exclusion Criteria:

* Anyone diagnosed with coronary heart disease, stroke, or cancer.
* Anyone with a severe disability who is unable to participate in the study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 150,000 adult China aged 35 to 74 who have lived in urban or rural areas of Fuzhou, Putian, Quanzhou, Nanping, Xiamen, Zhangzhou, Longyan, Sanming and Ningde in Fujian Province for more than 6 months without cardiovascular disease history and major disability.
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary Disease | 5 years
  It is a form of myocardial ischemia (insufficient blood supply to the heart muscle) caused by a decreased capacity of the coronary vessels. At the follow-up, the outcomes of coronary events were acquired. Coronary CTA examination and coronary angiography were the primary measuring modalities.

SECONDARY OUTCOMES:
other metabolic diseases | 5 years
  Including hypertension, stroke, diabetes, impaired glucose tolerance, obesity, cancer, chronic obstructive pulmonary disease and chronic kidney disease. These disorders were diagnosed using international standards, and the necessary information was gathered during face-to-face follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China